CLINICAL TRIAL: NCT01999972
Title: A PHASE 1B, OPEN LABEL, DOSE ESCALATION STUDY TO EVALUATE SAFETY, PHARMACOKINETICS AND PHARMACODYNAMICS OF AXITINIB (AG-013736) IN COMBINATION WITH CRIZOTINIB (PF-02341066) IN PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Phase 1b Study Of Axitinib In Combination With Crizotinib In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A4061068; 2015-001724-31 (EudraCT Number)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Advanced Solid Tumors
Keywords: Carcinoma; Renal Cell
MeSH Terms: conditions — Carcinoma | interventions — Axitinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Axitinib in combination with crizotinib, escalation phase (Experimental): Dose Escalation Advanced solid tumor that is resistant to standard therapy or for which no standard therapy is available
  Interventions: Drug: axitinib; Drug: crizotinib
- Expansion Phase Cohort 1 (Experimental): Dose Expansion, Cohort 1: axitinib in combination with crizotinib Advanced renal cell cancer [RCC] with no prior systemic therapy
  Interventions: Drug: axitinib; Drug: crizotinib
- Expansion Phase Cohort 2 (Experimental): Dose Expansion, Cohort 2: axitinib in combination with crizotinib Advanced renal cell cancer with at least one but no more than two prior systemic treatment regimens directed at advanced RCC
  Interventions: Drug: axitinib; Drug: crizotinib

INTERVENTIONS:
Drug: axitinib — Axitinib: tablets, dosage range 2 - 5 mg, given orally twice daily on a continuous dosing schedule in 28 days cycles.
  Arms: Axitinib in combination with crizotinib, escalation phase
Drug: crizotinib — Crizotinib: capsules, dosage range 200-250 mg, given orally twice daily or every day on a continuous dosing schedule in 28 days cycle.
  Arms: Axitinib in combination with crizotinib, escalation phase
Drug: axitinib — Axitinib: tablets, dosage be defined based on Arm 1 results, given orally twice daily on a continuous dosing schedule in 28 days cycles.
  Arms: Expansion Phase Cohort 1
Drug: crizotinib — Crizotinib: capsules, dosage be defined based on Arm 1 results, given orally twice daily or every day on a continuous dosing schedule in 28 days cycle.
  Arms: Expansion Phase Cohort 1
Drug: axitinib — Axitinib: tablets, dosage be defined based on Arm 1 results, given orally twice daily on a continuous dosing schedule in 28 days cycles.
  Arms: Expansion Phase Cohort 2
Drug: crizotinib — Crizotinib: capsules, dosage be defined based on Arm 1 results, given orally twice daily or every day on a continuous dosing schedule in 28 days cycle.
  Arms: Expansion Phase Cohort 2

SUMMARY:
Despite the success of anti-angiogenic therapy in multiple treatment settings, a fraction of patients are refractory to vascular endothelial growth factor (VEGF) inhibitor treatment, while the majority of patients will eventually develop evasive resistance. It is proposed that mesenchymal-epithelial transition factor (c-MET) and its ligand hepatocyte growth factor (HGF or scatter factor) contribute to VEGF inhibitor resistance, such that combining a c-MET inhibitor with a VEGF inhibitor will provide additional clinical activity compared to VEGF inhibitor alone. This hypothesis will be tested using the cMET/ALK inhibitor, crizotinib, in combination with the VEGF inhibitor, axitinib.Since this will be the first study of axitinib given in combination with crizotinib, the study will primarily assess the safety and tolerability of the combination regimen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis - Dose Escalation Phase: Histologically or cytologically confirmed diagnosis of advanced solid tumor that is resistant to standard therapy or for which no standard therapy is available.
* Diagnosis - Dose Expansion Phase: Histologically or cytologically confirmed advanced RCC with a component of clear cell subtype
* Dose Expansion Phase: at least one measureable lesion as defined by RECIST [Response Evaluation Criterion in Solid Tumors] version 1.1.
* ECOG [Eastern Cooperative Oncology Group] Performance Status 0 or 1.

Exclusion Criteria:

* Major surgery <4 weeks or radiation therapy <2 weeks of patient registration.
* History of or known active seizure disorder, brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
* Dose Expansion Phase only: diagnosis of any other malignancy within 2 years prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02-26 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (15):
  - University of Chicago Medical Center, Chicago, Illinois
  - Investigational Drug Services IUHSCC, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State University, Dept. of Oncology, Detroit, Michigan
  - University of Minnesota Health Clinics and Surgery Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview IDS Pharmacy, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - University of Minnesota Physicians Masonic Cancer Center, Minneapolis, Minnesota
  - Cleveland Clinic Taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - John A Moran Eye Center, Salt Lake City, Utah
  - University Station Ophthalmology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- United Kingdom (2):
  - St Bartholomew's Hospital - Barts Health NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Michaelson MD, Gupta S, Agarwal N, Szmulewitz R, Powles T, Pili R, Bruce JY, Vaishampayan U, Larkin J, Rosbrook B, Wang E, Murphy D, Wang P, Lechuga MJ, Valota O, Shepard DR. A Phase Ib Study of Axitinib in Combination with Crizotinib in Patients with Metastatic Renal Cell Cancer or Other Advanced Solid Tumors. Oncologist. 2019 Sep;24(9):1151-e817. doi: 10.1634/theoncologist.2018-0749. Epub 2019 Jun 6. PMID 31171735
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061068&StudyName=A%20Phase%201b%20Study%20Of%20Axitinib%20In%20Combination%20With%20Crizotinib%20In%20Patients%20With%20Advanced%20Solid%20Tumors%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 2 parts: Part 1 (Dose escalation part to determine maximum tolerated dose [MTD] of axitinib in combination with crizotinib), Part 2 (Dose expansion part to assess the safety and tolerability of axitinib in combination with crizotinib at MTD determined in Part 1).
Pre-assignment Details: To understand the pharmacokinetic (PK) effects of crizotinib on axitinib, a 7-day lead-in period of single-agent axitinib directly preceding the administration of the crizotinib and axitinib combination was included prior to Cycle 1 in the dose escalation phase of the study.
Groups:
- Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg: Participants received axitinib tablet at a dose of 3 milligrams (mg) orally, twice daily (BID) in combination with crizotinib capsule at a dose of 200 mg orally BID in each 28-day cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor.
- Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg: Participants received axitinib tablet at a dose of 3 mg orally BID in combination with crizotinib capsule at a dose of 250 mg orally BID in each 28-day cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor.
- Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg: Participants received axitinib tablet at a dose of 5 mg orally BID in combination with crizotinib capsule at a dose of 200 mg orally BID in each 28-day cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor.
- Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg: Participants received axitinib tablet at a dose of 5 mg orally BID in combination with crizotinib capsule at a dose of 250 mg orally BID in each 28-day cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor.
- Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg: Participants with advanced renal cell carcinoma (RCC) with no prior systemic therapy, received axitinib and crizotinib combination therapy at maximum tolerated dose (MTD) (axitinib tablet at a dose of 5 mg orally BID in combination with crizotinib capsule at a dose of 250 mg orally BID) in each 28-day cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor.
- Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg: Participants with advanced RCC with at least one but no more than two prior systemic therapy, received axitinib and crizotinib combination therapy at MTD (axitinib tablet at a dose of 5 mg orally BID in combination with crizotinib capsule at a dose of 250 mg orally BID) in each 28-day cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor.
Period: Dose Escalation Part
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Started | 5 | 3 | 5 | 11 | 0 | 0
Treated | 5 | 3 | 4 | 10 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 3 | 5 | 11 | 0 | 0
Not completed — Participant refused further follow-up | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Enrolled but not treated | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Disease progression | 3 | 2 | 3 | 6 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Global deterioration of health status | 1 | 0 | 0 | 1 | 0 | 0
Period: Dose Expansion Part
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Started | 0 | 0 | 0 | 0 | 21 | 7
Treated | 0 | 0 | 0 | 0 | 21 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 21 | 7
Not completed — Death | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Disease progression | 0 | 0 | 0 | 0 | 9 | 3
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Participant's non-compliance | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant refused further follow-up | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Changed to standard of care | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all enrolled participants who received at least 1 dose of axitinib or crizotinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg | Total
Number analyzed (Participants) | 5 | 3 | 4 | 10 | 21 | 7 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (2.2) | 48.7 (14.5) | 60.3 (6.2) | 63.9 (6.0) | 62.4 (7.9) | 61.9 (8.9) | 61.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5 | 6 | 0 | 16
  Male | 4 | 2 | 1 | 5 | 15 | 7 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 3 | 2 | 10 | 21 | 5 | 46
  Black | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose-Escalation Part: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: Toxicity as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03. DLT defined as any following events attributable to any (axitinib or crizotinib) or both agents in combination: hematologic (Grade 4 neutropenia, absolute neutrophil count<1000/mm^3 with single temperature of >38.3 degrees celsius or sustained temperature of 38 degrees celsius for >1 hour; >=Grade 3 neutropenic infection; >=Grade 3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia), non-hematologic (>=Grade 3 toxicities [except asymptomatic hypophosphatemia, hyperuricemia without signs, symptoms of gout, and tumor lysis syndrome], nausea, vomiting or diarrhea persisted at Grade 3 or 4 despite maximal medical therapy; Grade 3 hypertension if persistent despite anti-hypertensives); In asymptomatic participant, Grade 3 QTc prolongation (QTc>=501 msec) if persisted after correcting reversible causes, and failure to deliver >=75 percent (%) of dose of each study drug.
Time Frame: Cycle 1 (28 days)
Population: Per protocol analysis set:all enrolled participants who received at least 1 dose of study drug, experienced either DLT during first cycle,or completed first cycle observation period.Participants who lost to follow up before receiving at least 75% of planned first cycle dose due to reasons other than treatment-related AEs were not evaluable for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drugs (crizotinib and axitinib) without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and until 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: First dose of study drug until 28 days after last dose (up to 35 cycles in Part 1 and 35 cycles in Part 2, each cycle 28 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or crizotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 5 | 3 | 4 | 10 | 21 | 7
Participants
  AEs | 5 | 3 | 3 | 10 | 21 | 7
  SAEs | 2 | 2 | 0 | 5 | 8 | 3

3. Secondary Outcome: Number of Participants With Treatment-Related Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drugs (crizotinib and axitinib) in a participant who received study drugs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and until 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: as for outcome 2
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or crizotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 5 | 3 | 4 | 10 | 21 | 7
Participants
  AEs | 4 | 3 | 3 | 9 | 21 | 6
  SAEs | 1 | 0 | 0 | 2 | 1 | 2

4. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events (AEs) as Graded by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.03
Description: An AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Grade 3 (severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death. Grade 5 = death. Treatment-emergent were events between first dose of study drug and until 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: as for outcome 2
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or crizotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 5 | 3 | 4 | 10 | 21 | 7
Participants
  Grade 3 or 4 AEs | 3 | 3 | 1 | 8 | 19 | 6
  Grade 5 AEs | 0 | 1 | 0 | 0 | 2 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.03: Hematological Test Abnormalities
Description: Laboratory parameters included hematological and biochemistry parameters. Hematological parameters included haemoglobin (anemia, haemoglobin increased), lymphocytes (lymphopenia, lymphocyte count increased), neutrophils, platelets and white blood cells. Number of participants with hematological abnormalities by grades (as per NCI CTCAE version 4.03) were reported. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: Baseline up to end of treatment (up to 35 cycles in Part 1 and 35 cycles in Part 2, each cycle 28 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or crizotinib. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 21 | 6
Participants
  Anemia: Grade 1 | 1 | 1 | 0 | 2 | 10 | 3
  Anemia: Grade 2 | 0 | 0 | 0 | 1 | 2 | 2
  Anemia: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0
  Anemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 | 0 | 1 | 0 | 1 | 1 | 0
  Hemoglobin increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphopenia: Grade 1 | 1 | 0 | 0 | 1 | 0 | 0
  Lymphopenia: Grade 2 | 0 | 0 | 1 | 2 | 7 | 4
  Lymphopenia: Grade 3 | 1 | 0 | 0 | 2 | 2 | 0
  Lymphopenia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (absolute): Grade 1 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophils (absolute): Grade 2 | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophils (absolute): Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (absolute): : Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 1 | 0 | 1 | 1 | 2 | 6 | 2
  Platelets: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cells: Grade 1 | 1 | 0 | 1 | 0 | 6 | 1
  White blood cells: Grade 2 | 0 | 0 | 0 | 0 | 1 | 1
  White blood cells: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cells: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.03: Biochemistry Test Abnormalities
Description: Laboratory parameters included hematological and biochemistry parameters. Biochemistry parameters/abnormalities included alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, bilirubin (total), creatinine, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia and gamma glutamyl transferase Number of participants with biochemistry test abnormalities by grades (NCI CTCAE version 4.03) were reported. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: Baseline up to end of treatment (up to 35 cycles in Part 1 and 35 cycles in Part 2, each cycle 28 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or crizotinib. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 21 | 6
Participants
  Alanine aminotransferase: Grade 1 | 1 | 1 | 2 | 3 | 6 | 1
  Alanine aminotransferase: Grade 2 | 0 | 0 | 1 | 1 | 3 | 0
  Alanine aminotransferase: Grade 3 | 0 | 1 | 0 | 1 | 2 | 0
  Alanine aminotransferase: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase: Grade 1 | 1 | 1 | 3 | 6 | 9 | 0
  Alkaline phosphatase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase: Grade 1 | 1 | 1 | 3 | 3 | 7 | 2
  Aspartate aminotransferase: Grade 2 | 0 | 0 | 0 | 2 | 3 | 0
  Aspartate aminotransferase: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0
  Aspartate aminotransferase: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (total): Grade 1 | 0 | 0 | 0 | 0 | 1 | 0
  Bilirubin (total): Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (total): Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (total): Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Grade 1 | 3 | 1 | 2 | 8 | 16 | 2
  Creatinine: Grade 2 | 0 | 1 | 1 | 0 | 3 | 2
  Creatinine: Grade 3 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 1 | 0 | 0 | 0 | 0 | 2 | 1
  Hypercalcemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia: Grade 1 | 2 | 1 | 3 | 4 | 13 | 3
  Hyperglycemia: Grade 2 | 0 | 0 | 0 | 4 | 5 | 1
  Hyperglycemia: Grade 3 | 0 | 1 | 0 | 0 | 1 | 0
  Hyperglycemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1 | 0 | 0 | 1 | 1 | 5 | 0
  Hyperkalemia: Grade 2 | 0 | 0 | 0 | 0 | 1 | 0
  Hyperkalemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 | 0 | 0 | 1 | 1 | 3 | 1
  Hypermagnesemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 1 | 0 | 0 | 0 | 0 | 1 | 0
  Hypernatremia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 | 2 | 2 | 0 | 1 | 3 | 0
  Hypoalbuminemia: Grade 2 | 0 | 0 | 1 | 3 | 6 | 4
  Hypoalbuminemia: Grade 3 | 0 | 0 | 0 | 0 | 2 | 0
  Hypoalbuminemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 1 | 0 | 0 | 1 | 1 | 9 | 2
  Hypocalcemia: Grade 2 | 0 | 0 | 0 | 0 | 2 | 1
  Hypocalcemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 1 | 0 | 0 | 0 | 0 | 4 | 0
  Hypoglycemia: Grade 2 | 0 | 0 | 0 | 0 | 2 | 0
  Hypoglycemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1 | 0 | 0 | 0 | 0 | 1 | 0
  Hypokalemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 3 | 0 | 0 | 2 | 0 | 0 | 0
  Hypokalemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 | 0 | 0 | 2 | 0 | 2 | 1
  Hypomagnesemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 1 | 0 | 1 | 0 | 2 | 5 | 1
  Hyponatremia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 | 0 | 0 | 0 | 1 | 0 | 0
  Hyponatremia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia: Grade 2 | 0 | 1 | 1 | 4 | 6 | 3
  Hypophosphatemia: Grade 3 | 0 | 0 | 0 | 1 | 5 | 1
  Hypophosphatemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma glutamyl transferase : Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Gamma glutamyl transferase : Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma glutamyl transferase : Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Gamma glutamyl transferase : Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma glutamyl transferase : Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Gamma glutamyl transferase : Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma glutamyl transferase : Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Gamma glutamyl transferase : Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Day 1, 15 of Cycle 1, Day 1 of Cycles 2, 4, 6, 12, 24 and End of Treatment Visit
Time Frame: Baseline; Day 1 and 15 of Cycle 1; Day 1 of Cycles 2, 4, 6, 12, 24; and end of treatment (up to a maximum duration of 35 cycles in Part 1 and 35 cycles in Part 2, each cycle 28 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or crizotinib. Here, '0' in the "number analyzed" field signifies that none of the participant were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 5 | 3 | 4 | 10 | 21 | 7
millimeters of mercury (mmHg)
  SBP: At Baseline | 115.7 (13.66) | 116.2 (4.91) | 124.8 (9.17) | 113.6 (12.16) | 131.4 (15.58) | 139.7 (14.41)
  SBP: Change at Cycle 1 Day 1: number analyzed (Participants) | 4 | 3 | 3 | 10 | 11 | 0
  SBP: Change at Cycle 1 Day 1 | 2.0 (7.25) | 17.3 (2.25) | 14.5 (14.76) | 15.5 (14.92) | -1.7 (19.34) |
  SBP: Change at Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 8 | 21 | 4
  SBP: Change at Cycle 1 Day 15 | 6.8 (9.00) | 3.5 (10.04) | 8.7 (9.45) | 12.0 (18.21) | 4.2 (17.06) | -1.9 (9.47)
  SBP: Change at Cycle 2 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 7 | 21 | 5
  SBP: Change at Cycle 2 Day 1 | 0.7 (8.13) | 4.3 (3.33) | 0.7 (9.81) | 0.9 (7.47) | -1.8 (10.40) | -11.5 (20.04)
  SBP: Change at Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 6 | 18 | 5
  SBP: Change at Cycle 4 Day 1 |  | 3.5 | -5.8 (8.01) | 2.3 (17.01) | -0.4 (12.75) | -14.2 (7.54)
  SBP: Change at Cycle 6 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 3 | 15 | 5
  SBP: Change at Cycle 6 Day 1 |  | -15.0 | 9.8 (19.45) | 1.5 (15.90) | 0.3 (18.57) | -10.4 (17.50)
  SBP: Change at Cycle 12 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 2 | 6 | 2
  SBP: Change at Cycle 12 Day 1 |  | -7.5 | -7.0 | -7.3 (1.77) | -5.8 (14.54) | -14.0 (2.83)
  SBP: Change at Cycle 24 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 0
  SBP: Change at Cycle 24 Day 1 |  |  | 7.0 | 9.0 | -9.0 |
  SBP: End of Treatment: number analyzed (Participants) | 3 | 2 | 3 | 7 | 19 | 6
  SBP: End of Treatment | -7.0 (13.44) | -4.8 (10.25) | -14.0 (17.58) | 4.9 (9.32) | -0.7 (15.17) | -12.4 (22.00)
  DBP: At Baseline | 76.8 (11.99) | 83.0 (4.77) | 83.5 (3.03) | 75.8 (7.66) | 78.5 (10.59) | 76.7 (10.37)
  DBP: Change at Cycle 1 Day 1: number analyzed (Participants) | 4 | 3 | 3 | 10 | 11 | 0
  DBP: Change at Cycle 1 Day 1 | 2.1 (4.57) | 4.2 (7.77) | 4.8 (5.30) | 7.0 (11.23) | 5.3 (8.84) |
  DBP: Change at Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 8 | 21 | 4
  DBP: Change at Cycle 1 Day 15 | 0.7 (12.34) | -2.2 (1.04) | 2.5 (11.65) | 3.9 (8.51) | 1.8 (10.43) | -7.5 (10.54)
  DBP: Change at Cycle 2 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 7 | 21 | 5
  DBP: Change at Cycle 2 Day 1 | -2.8 (7.09) | -2.3 (2.57) | 0.5 (3.12) | -2.3 (5.61) | 0.5 (8.36) | -2.4 (6.01)
  DBP: Change at Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 6 | 18 | 5
  DBP: Change at Cycle 4 Day 1 |  | 3.0 | -4.8 (2.02) | -2.6 (7.94) | -1.0 (10.24) | -4.7 (4.89)
  DBP: Change at Cycle 6 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 3 | 15 | 5
  DBP: Change at Cycle 6 Day 1 |  | -17.5 | -0.5 (14.14) | -6.0 (4.92) | -3.0 (13.62) | -1.4 (12.96)
  DBP: Change at Cycle 12 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 2 | 6 | 2
  DBP: Change at Cycle 12 Day 1 |  | -7.0 | 2.5 | -7.5 (7.07) | -0.3 (11.25) | -5.5 (1.41)
  DBP: Change at Cycle 24 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 0
  DBP: Change at Cycle 24 Day 1 |  |  | -1.0 | 7.0 | -6.5 |
  DBP: End of Treatment: number analyzed (Participants) | 3 | 2 | 3 | 7 | 19 | 6
  DBP: End of Treatment | -1.5 (4.44) | -4.5 (4.24) | -6.2 (8.13) | -2.3 (9.58) | -2.8 (10.94) | -4.8 (11.17)

8. Secondary Outcome: Change From Baseline in Pulse Rate at Day 1, 15 of Cycle 1, Day 1 of Cycles 2, 4, 6, 12, 24 and End of Treatment
Time Frame: Baseline; Day 1 and 15 of Cycle 1; Day 1 of Cycles 2, 4, 6, 12, 24; and end of treatment (any time up to a maximum duration of 35 cycles in Part 1 and 35 cycles in Part 2, each cycle 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 5 | 3 | 4 | 10 | 21 | 7
beats per minute (bpm)
  Pulse Rate: At Baseline | 88.4 (21.76) | 81.2 (4.25) | 82.6 (15.05) | 80.9 (7.70) | 73.9 (14.71) | 77.4 (11.66)
  Pulse Rate: Change at Cycle 1 Day 1: number analyzed (Participants) | 4 | 3 | 3 | 10 | 11 | 0
  Pulse Rate: Change at Cycle 1 Day 1 | -0.6 (9.44) | 5.3 (9.29) | -7.8 (1.44) | -0.3 (9.15) | -0.0 (12.25) |
  Pulse Rate: Change at Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 8 | 21 | 4
  Pulse Rate: Change at Cycle 1 Day 15 | -16.0 (7.26) | -12.7 (6.33) | -7.7 (26.63) | -8.1 (9.20) | -3.8 (11.55) | -14.1 (11.93)
  Pulse Rate: Change at Cycle 2 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 7 | 21 | 5
  Pulse Rate: Change at Cycle 2 Day 1 | -10.8 (15.25) | -1.5 (6.14) | -8.2 (23.91) | -0.4 (12.09) | -7.5 (11.39) | -15.3 (13.26)
  Pulse Rate: Change at Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 6 | 18 | 5
  Pulse Rate: Change at Cycle 4 Day 1 |  | -4.0 | -9.7 (4.54) | -3.7 (8.45) | -0.4 (16.15) | -11.1 (7.97)
  Pulse Rate: Change at Cycle 6 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 3 | 15 | 5
  Pulse Rate: Change at Cycle 6 Day 1 |  | -7.0 | -7.5 (7.78) | -8.5 (13.31) | -4.7 (18.60) | -3.1 (23.69)
  Pulse Rate: Change at Cycle 12 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 2 | 6 | 2
  Pulse Rate: Change at Cycle 12 Day 1 |  | 1.0 | 10.0 | -4.8 (6.72) | -2.8 (9.75) | -2.5 (7.78)
  Pulse Rate: Change at Cycle 24 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 0
  Pulse Rate: Change at Cycle 24 Day 1 |  |  | -11.0 | -20.5 | 2.0 |
  Pulse Rate: Change at End of Treatment: number analyzed (Participants) | 3 | 2 | 3 | 7 | 19 | 6
  Pulse Rate: Change at End of Treatment | -19.3 (11.59) | 8.0 (12.73) | -2.8 (12.89) | -1.2 (11.55) | 5.4 (20.42) | 17.6 (18.80)

9. Secondary Outcome: Change From Baseline in Body Weight at Day 1, 15 of Cycle 1, Day 1 of Cycles 2, 4, 6, 12, 24 and End of Treatment
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 5 | 3 | 4 | 10 | 21 | 7
kilograms
  Body Weight: At Baseline | 74.96 (11.339) | 87.43 (9.684) | 78.46 (13.938) | 82.63 (18.346) | 86.54 (17.044) | 93.00 (17.820)
  Body Weight: Change at Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 8 | 9 | 0
  Body Weight: Change at Cycle 1 Day 1 | -1.03 (0.379) | -1.43 (0.751) | -1.51 (1.917) | -0.98 (0.829) | -0.63 (2.227) |
  Body Weight: Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 8 | 21 | 4
  Body Weight: Cycle 1 Day 15 | -1.17 (1.747) | -3.87 (2.003) | -2.40 (3.064) | -1.56 (1.565) | -1.16 (2.305) | -1.72 (1.648)
  Body Weight: Change at Cycle 2 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 7 | 21 | 5
  Body Weight: Change at Cycle 2 Day 1 | -2.08 (3.123) | -6.27 (2.403) | -3.92 (3.806) | -2.28 (2.689) | -2.04 (3.109) | -1.21 (3.734)
  Body Weight: Change at Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 6 | 18 | 5
  Body Weight: Change at Cycle 4 Day 1 |  | -2.60 | -5.77 (5.228) | -3.36 (2.783) | -4.22 (4.118) | -2.80 (3.609)
  Body Weight: Change at Cycle 6 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 3 | 15 | 5
  Body Weight: Change at Cycle 6 Day 1 |  | -3.63 | -14.06 | -3.82 (5.538) | -4.18 (5.232) | -4.57 (6.264)
  Body Weight: Change at Cycle 12 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 2 | 6 | 2
  Body Weight: Change at Cycle 12 Day 1 |  | -4.20 | -11.40 | 2.11 (2.786) | -3.53 (4.366) | -6.15 (5.162)
  Body Weight: Change at Cycle 24 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 0
  Body Weight: Change at Cycle 24 Day 1 |  |  | -16.50 | 8.16 | -2.40 |
  Body Weight: Change at End of Treatment: number analyzed (Participants) | 3 | 2 | 3 | 6 | 19 | 5
  Body Weight: Change at End of Treatment | -2.17 (5.327) | -6.45 (6.576) | -13.60 (7.400) | -2.05 (7.134) | -5.46 (5.505) | -10.68 (9.058)

10. Secondary Outcome: Number of Participants With Change From Baseline in Eastern Cooperative Oncology Group Performance Status (ECOG-PS) to Worst Value
Description: ECOG-PS: used to assess how disease affected the daily living abilities of participant. It ranges on the scale from: 0-5 (0=fully active/able to carry on all pre-disease activities without restriction;1=restricted in physically strenuous activity but ambulatory/able to carry out light/sedentary work;2=ambulatory [for more than (>)50%of waking hours], capable of all self-care but unable to carry out any work activities;3=capable of limited self-care, confined to bed or chair [for >50% of waking hours];4=completely disabled, not capable of any self-care, totally confined to bed or chair;5= dead, higher score=more functional impairment) and changes to worst status scores were presented. Baseline value=value collected prior to first dose of study drug on Cycle 1 Day 1. Worst post-baseline value=worst value between first dose of any study drug and end of treatment (EOT) visit. Shift to low refers to lower than Baseline value; shift to high refers to higher than baseline value for ECOG-PS.
Time Frame: Baseline, End of Treatment (up to Cycle 35 [for Part 1] and up to Cycle 35 [for Part 2], each cycle 28 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or crizotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 5 | 3 | 4 | 10 | 21 | 7
Participants
  Baseline 0, EOT 0 | 0 | 0 | 0 | 0 | 3 | 1
  Baseline 0, EOT 1 | 1 | 1 | 2 | 1 | 8 | 0
  Baseline 0, EOT 2 | 0 | 0 | 0 | 2 | 0 | 0
  Baseline 0, EOT 3 | 0 | 0 | 0 | 1 | 0 | 0
  Baseline 0, EOT 4 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 1, EOT 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 1, EOT 1 | 3 | 1 | 0 | 6 | 7 | 2
  Baseline 1, EOT 2 | 1 | 0 | 1 | 0 | 2 | 2
  Baseline 1, EOT 3 | 0 | 1 | 0 | 0 | 1 | 0
  Baseline 1, EOT 4 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 2, EOT 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 2, EOT 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 2, EOT 2 | 0 | 0 | 0 | 0 | 0 | 1
  Baseline 2, EOT 3 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 2, EOT 4 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 3, EOT 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 3, EOT 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 3, EOT 2 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 3, EOT 3 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 3, EOT 4 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 4, EOT 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 4, EOT 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 4, EOT 2 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 4, EOT 3 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline 4, EOT 4 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Maximum Increase From Baseline in QTc Interval
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR) and by Bazette's formula (QTcB = QT divided by square root of RR). Number of participants with maximum increase from baseline of less than (<) 30 milliseconds (msec), 30 to <60 msec and greater than or equal to (>=) 60 msec were reported.
Time Frame: Baseline, End of Treatment (up to Cycle 35 [for Part 1] and up to Cycle 35 [for Part 2], each cycle 28 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or crizotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 5 | 3 | 4 | 10 | 21 | 7
Participants
  QTcF (msec): <30 | 2 | 1 | 2 | 8 | 16 | 4
  QTcF (msec): 30-60 | 2 | 2 | 0 | 1 | 4 | 2
  QTcF (msec): >=60 | 0 | 0 | 0 | 1 | 0 | 0
  QTcB (msec): <30 | 3 | 1 | 1 | 8 | 15 | 4
  QTcB (msec): 30 - 60 | 1 | 2 | 1 | 1 | 5 | 2
  QTcB (msec): >=60 | 0 | 0 | 0 | 1 | 0 | 0

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Axitinib and Crizotinib
Description: Data of this outcome measure was not planned to be analyzed for Cohort 2 in dose expansion part, as pre-specified in protocol.
Time Frame: Axitinib: Pre-dose (0 hour [hr]), 1, 2, 3, 4, 6, 8 hrs post-dose at Lead-in Day 7, Cycle 1 Day 15; Crizotinib: pre-dose (0 hr), 1, 2, 3, 4, 6, 8 hrs post-dose at Cycle 1 Day 15
Population: Pharmacokinetic (PK) parameter analysis population was defined as all treated participants who had at least 1 of the PK parameters of interest of any of the study drugs.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 4 | 3 | 3 | 10 | 12
nanogram per milliliter
  Axitinib: Lead-in Day 7: number analyzed (Participants) | 2 | 3 | 2 | 4 | 7
  Axitinib: Lead-in Day 7 | 8.777 (34) | 21.33 (12) | 31.31 (31) | 25.32 (101) | 40.21 (34)
  Axitinib: Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 2 | 4 | 7
  Axitinib: Cycle 1 Day 15 | 6.532 (55) | 24.28 (115) | 30.89 (33) | 25.02 (77) | 40.91 (55)
  Crizotinib: Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 2 | 6 | 7
  Crizotinib: Cycle 1 Day 15 | 194.8 (6) | 230.8 (35) | 169.9 (298) | 207.0 (43) | 235.9 (99)

13. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Axitinib and Crizotinib
Description: as for outcome 12
Time Frame: as for outcome 12
Population: The PK parameter analysis population was defined as all treated participants who had at least 1 of the PK parameters of interest of any of the study drugs.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 4 | 3 | 3 | 10 | 12
hours
  Axitinib: Lead-in Day 7: number analyzed (Participants) | 2 | 3 | 2 | 4 | 7
  Axitinib: Lead-in Day 7 | 2.09 [2.03 to 2.15] | 2.00 [1.03 to 2.00] | 2.48 [1.95 to 3.00] | 3.49 [1.00 to 4.00] | 2.00 [1.00 to 3.98]
  Axitinib: Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 2 | 4 | 7
  Axitinib: Cycle 1 Day 15 | 1.50 [1.00 to 2.00] | 3.00 [3.00 to 6.00] | 1.50 [1.00 to 2.00] | 1.50 [1.00 to 2.00] | 2.00 [1.00 to 3.00]
  Crizotinib: Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 2 | 6 | 7
  Crizotinib: Cycle 1 Day 15 | 12.00 [12.00 to 12.00] | 3.92 [3.07 to 6.00] | 7.00 [2.00 to 12.00] | 3.00 [1.00 to 8.00] | 3.22 [1.00 to 8.08]

14. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Axitinib and Crizotinib
Description: Area under the plasma concentration versus time-curve from time zero to end of dosing interval (AUCtau), where dosing interval was 12 hours. Data of this outcome measure was not planned to be analyzed for Cohort 2 in dose expansion part, as pre-specified in protocol.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 4 | 3 | 3 | 10 | 12
nanogram*hour per milliliter
  Axitinib: Lead-in Day 7: number analyzed (Participants) | 2 | 3 | 2 | 3 | 7
  Axitinib: Lead-in Day 7 | 31.96 (61) | 105.9 (29) | 131.6 (149) | 93.22 (135) | 197.8 (46)
  Axitinib: Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 2 | 3 | 7
  Axitinib: Cycle 1 Day 15 | 34.87 (65) | 143.8 (107) | 196.8 (6) | 127.4 (121) | 208.6 (35)
  Crizotinib: Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 2 | 6 | 7
  Crizotinib: Cycle 1 Day 15 | 1905 (10) | 2162 (33) | 1526 (316) | 1985 (41) | 2144 (105)

15. Secondary Outcome: Apparent Oral Clearance (CL/F) of Axitinib and Crizotinib
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent oral clearance was obtained by dividing study drug dose with AUCtau, where AUCtau was area under the plasma concentration-time curve from time zero to the quantifiable concentration at the end of dosing interval. Data of this outcome measure was not planned to be analyzed for Cohort 2 in dose expansion part, as pre-specified in protocol.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 4 | 3 | 3 | 10 | 12
liters per hour
  Axitinib: Lead-in Day 7: number analyzed (Participants) | 2 | 3 | 2 | 3 | 7
  Axitinib: Lead-in Day 7 | 94.06 (61) | 28.32 (29) | 38.03 (149) | 53.70 (134) | 25.32 (46)
  Axitinib: Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 2 | 3 | 7
  Axitinib: Cycle 1 Day 15 | 86.03 (65) | 20.86 (107) | 25.38 (6) | 39.28 (121) | 23.96 (35)
  Crizotinib: Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 2 | 6 | 7
  Crizotinib: Cycle 1 Day 15 | 105.0 (10) | 115.7 (33) | 131.2 (316) | 126.0 (41) | 116.6 (105)

16. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Axitinib and Crizotinib
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 12
Population: Data for this outcome measure was not collected due to change in planned analysis.
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based on assessment of confirmed complete response [CR] or confirmed partial response [PR] according to Response Evaluation Criteria In Solid Tumors [RECIST] version1.1 were reported. Confirmed responses were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as disappearance of all lesions (target and/or non target). PR were those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent.
Time Frame: From Baseline until disease progression or death, whichever occurred first (up to 35 cycles in Part 1 and 35 cycles in Part 2, each cycle 28 days)
Population: Response-evaluable analysis set included all participants who received at least 1 dose of axitinib and crizotinib and had an adequate baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 4 | 3 | 3 | 9 | 20 | 7
percentage of participants | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 33.6] | 40.0 [19.1 to 63.9] | 14.3 [0.4 to 57.9]

18. Secondary Outcome: Dose Expansion Part: Duration of Response
Description: Duration of response (as per Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) was defined as the time (in months) from first documentation of objective tumor response (complete response [CR] or partial response [PR]) until the first date that recurrent, progressive disease, or death (whichever occurred first). CR was defined as disappearance of all lesions (target and/or non target). PR were those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent. Progression was defined as >= 20 percent increase in sum of longest diameter of target lesions; measurable increase in non-target lesion; appearance of new lesions.
Time Frame: From first objective response until first recurrent, disease progression, or death, whichever occurred first (up to 35 cycles, each cycle 28 days)
Population: Subset of response evaluable analysis set included all participants with overall objective response of CR or PR who received at least 1 dose of axitinib and crizotinib and had baseline tumor assessment. Data for this outcome measure was not planned to be collected and analyzed for "dose escalation part", as pre specified in protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 8 | 1
months | 9.7 [3.6 to 28.6] | NA [NA to NA] — Data not estimable due to small number of participants with an event.

19. Secondary Outcome: Dose Expansion Part: Progression-Free Survival (PFS)
Description: PFS (as per Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) was defined as the time (in months) from start of study treatment to first documentation of objective tumor progression or death due to any cause, whichever occurred first. PFS (in months) was calculated as (first event date minus date of first dose of study medication plus 1) divided by 30.44. Progression was defined as >= 20 percent increase in sum of longest diameter of target lesions; measurable increase in non-target lesion; appearance of new lesions. PFS was not estimated in Dose Expansion Cohort 2 due to small sample size.
Time Frame: From Baseline until disease progression or death, whichever occurred first (up to 35 cycles, each cycle 28 days)
Population: Response-evaluable analysis set included all participants who received at least 1 dose of axitinib and crizotinib and had an adequate baseline tumor assessment. Data for this outcome measure was not planned to be collected and analyzed for "dose escalation part", as pre specified in protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 20 | 7
months | 5.6 [3.5 to 13.6] | NA [NA to NA] — Data not estimable due to small number of participants with an event.

20. Secondary Outcome: Dose Expansion Part Cohort 1: Levels of Serum Soluble Protein Biomarkers
Description: Serum soluble protein biomarkers included angiopoietin-2, Hepatocyte Growth Factor (HGF), Vascular Endothelial Growth Factor Receptor 3 (VEGFR 3). Biomarker analysis was not planned to be performed in dose escalation part and Cohort 2 of dose expansion part, as pre-specified in protocol.
Time Frame: Baseline, Cycle 2 Day 1, end of treatment (up to 35 cycles, each cycle 28 days)
Population: Serum soluble protein biomarker analysis set included all enrolled participants who received at least one dose of any study drug, and had at least one biomarker parameter from the corresponding assay sample with at least one baseline biomarker measurement.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 19
nanograms per milliliter (ng/mL)
  Angiopoietin-2: Baseline | 4.84 (5.282)
  Angiopoietin-2: Cycle 2 Day 1: number analyzed (Participants) | 18
  Angiopoietin-2: Cycle 2 Day 1 | 3.81 (2.351)
  Angiopoietin-2: End of Treatment: number analyzed (Participants) | 8
  Angiopoietin-2: End of Treatment | 5.44 (2.996)
  HGF: Baseline | 9.59 (4.831)
  HGF: Cycle 2 Day 1: number analyzed (Participants) | 18
  HGF: Cycle 2 Day 1 | 15.58 (22.897)
  HGF: End of Treatment: number analyzed (Participants) | 8
  HGF: End of Treatment | 11.95 (5.237)
  VEGFR3: Baseline | 35.368 (8.6166)
  VEGFR3: Cycle 2 Day 1: number analyzed (Participants) | 18
  VEGFR3: Cycle 2 Day 1 | 26.000 (8.3314)
  VEGFR3: End of Treatment: number analyzed (Participants) | 8
  VEGFR3: End of Treatment | 36.444 (20.2426)

21. Secondary Outcome: Dose Expansion Part Cohort 1: Change From Baseline in Serum Concentration of Circulating microRNAs (miRNA) at End of Treatment
Time Frame: Baseline, end of treatment (up to 35 cycles, each cycle 28 days)
Population: This outcome measure was not analyzed because of a change in planned analysis, due to the lack of strong evidence available supporting testing a hypothesis in the small sample set.
Arm/Group | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 0

22. Secondary Outcome: Dose Expansion Part Cohort 1: Percentage of c-MET Positive Tumor Cell at Baseline in Relation to Objective Response Rate (ORR)
Description: Percentage of c-MET positive tumor cell for objective response (complete response [CR] + partial response [PR]) is reported. Objective response was defined as CR and PR. CR was defined as disappearance of all lesions (target and/or non target). PR were those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent. Biomarker analysis was not planned to be performed in dose escalation part and Cohort 2 of dose expansion part, as pre-specified in protocol.
Time Frame: Baseline
Population: Tumor Immunohistochemistry (IHC) analysis set included all enrolled participants who received at least one dose of any study drug, and had at least one biomarker parameter from the corresponding assay sample with at least one baseline biomarker measurement, and had confirmed objective response (CR+PR).
Measure: Mean (Standard Deviation); unit: percentage of positive tumor cells
Arm/Group | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 5
percentage of positive tumor cells
  Percent positive cell c-MET Cytoplasmic: CR +PR | 70.0 (25.50)
  Percent positive cell c-MET Membrane: CR + PR | 85.0 (20.62)

23. Secondary Outcome: Dose Expansion Part Cohort 1: Level of Plasma Soluble Protein Biomarker (c-MET)
Description: Plasma soluble protein biomarker included c-MET. Biomarker analysis was not planned to be performed in dose escalation part and Cohort 2 of dose expansion part, as pre-specified in protocol.
Time Frame: Baseline; Day 1 and 15 of Cycle 1; Day 1 of Cycles 2, 3, 5; end of treatment (up to 35 cycles, each cycle 28 days)
Population: Plasma soluble protein biomarker analysis set included all enrolled participants who received at least one dose of any study drug, and had at least one biomarker parameter from the corresponding assay sample with at least one baseline biomarker measurement.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 19
nanogram per milliliter (ng/mL)
  c-MET: Baseline | 640.0 (120.77)
  c-MET: Cycle 1 Day 1: number analyzed (Participants) | 11
  c-MET: Cycle 1 Day 1 | 667.4 (117.09)
  c-MET: Cycle 1 Day 15: number analyzed (Participants) | 17
  c-MET: Cycle 1 Day 15 | 694.8 (143.41)
  c-MET: Cycle 2 Day 1: number analyzed (Participants) | 18
  c-MET: Cycle 2 Day 1 | 757.1 (148.75)
  c-MET: Cycle 3 Day 1: number analyzed (Participants) | 17
  c-MET: Cycle 3 Day 1 | 678.2 (120.46)
  c-MET: Cycle 5 Day 1: number analyzed (Participants) | 16
  c-MET: Cycle 5 Day 1 | 689.8 (158.09)
  c-MET: End of Treatment: number analyzed (Participants) | 7
  c-MET: End of Treatment | 759.0 (183.74)

24. Secondary Outcome: Dose Expansion Part Cohort 1: Ratio of Serum Soluble Protein Biomarkers Level to Baseline Biomarkers Level by Each Timepoint
Description: Serum soluble protein biomarkers included angiopoietin-2, Hepatocyte Growth Factor (HGF), Vascular Endothelial Growth Factor Receptor 3 (VEGFR3). Ratio=value of serum soluble protein biomarkers at each time point to the value at baseline. Biomarker analysis was not planned to be performed in dose escalation part and Cohort 2 of dose expansion part, as pre-specified in protocol.
Time Frame: Baseline, Cycle 2 Day 1, end of treatment (up to 35 cycles, each cycle 28 days)
Population: Serum soluble protein biomarker analysis set: all enrolled participants who received at least 1 dose of any study drug, had at least 1 biomarker parameter from corresponding assay sample with at least 1 baseline biomarker measurement. Here, 'number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg
Number analyzed (Participants) | 18
ratio
  Angiopoietin-2- (Cycle 2 Day 1 ratio Baseline) | 0.90 (0.321)
  Angiopoietin-2 (End of Treatment ratio Baseline): number analyzed (Participants) | 8
  Angiopoietin-2 (End of Treatment ratio Baseline) | 1.50 (1.056)
  HGF (Cycle 2 Day 1 ratio Baseline) | 1.62 (1.449)
  HGF (End of Treatment ratio Baseline): number analyzed (Participants) | 8
  HGF (End of Treatment ratio Baseline) | 1.18 (0.278)
  VEGFR3 (Cycle 2 Day 1 ratio Baseline) | 0.748 (0.1869)
  VEGFR3 (End of Treatment ratio Baseline): number analyzed (Participants) | 8
  VEGFR3 (End of Treatment ratio Baseline) | 0.969 (0.6246)

ADVERSE EVENTS:
Time Frame: Baseline up to end of treatment (up to 35 cycles in Part 1 and 35 cycles in Part 2, each cycle 28 days)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/3 | 0/4 | 0/10 | 2/21 | 1/7
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/3 | 0/4 | 5/10 | 8/21 | 3/7
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 3/4 | 10/10 | 21/21 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg (N=5) | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg (N=3) | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg (N=4) | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg (N=10) | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg (N=21) | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg (N=7)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dose Escalation Part: Crizotinib 200mg+Axitinib 3mg (N=5) | Dose Escalation Part: Crizotinib 250mg+Axitinib 3mg (N=3) | Dose Escalation Part: Crizotinib 200 mg+Axitinib 5 mg (N=4) | Dose Escalation Part: Crizotinib 250 mg+Axitinib 5 mg (N=10) | Dose Expansion Part: Cohort 1 Crizotinib 250 mg+Axitinib 5 mg (N=21) | Dose Expansion Part: Cohort 2 Crizotinib 250 mg+Axitinib 5 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 2 | 2 | 1 | 3 | 0
Eyelid pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3 | 6 | 16 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 6 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 7 | 19 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 2 | 5 | 12 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Tongue discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 3 | 7 | 9 | 5
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 3 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 3 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 7 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 1 | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 0 | 3 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 3 | 8 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 3
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 3 | 5 | 7 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 6 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 3 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 4 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 4 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 2 | 3 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 3 | 2 | 0 | 3 | 5 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 4 | 11 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1/2 | 0 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 3 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 2 | 2 | 4 | 7 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 3 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-01-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT01999972/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT01999972/SAP_001.pdf